CLINICAL TRIAL: NCT01097330
Title: Catheter Ablation Versus Amiodarone for Shock Prophylaxis in Defibrillator Patients With Ventricular Tachycardia: A Multi-center Randomized Trial
Brief Title: Catheter Ablation Versus Amiodarone for Shock Prophylaxis in Defibrillator Patients With Ventricular Tachycardia
Acronym: CEASE-VT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Anticipated non-feasibility of recruitment objectives
Sponsor: Population Health Research Institute (Other)
Collaborators: Abbott Medical Devices (Industry); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEASE-VT
Record Dates: First submitted 2010-03-31; First posted 2010-04-01 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Defibrillators, Implantable; Tachycardia, Ventricular
Keywords: Defibrillators, Implantable; Tachycardia, Ventricular; Catheter Ablation; Amiodarone
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Catheter Ablation; Radiofrequency Ablation; Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ablation (Active Comparator): Catheter based radiofrequency ablation for ischemic ventricular tachycardia
  Interventions: Procedure: Ablation
- Amiodarone (Active Comparator): amiodarone titrated to therapeutic levels as per standard of care and maintained on a dose of at least 200 mg (300 mg recommended) once a day for the duration of the study.
  Interventions: Drug: Amiodarone

INTERVENTIONS:
Procedure: Ablation — Catheter based radiofrequency ablation for ischemic ventricular tachycardia scheduled to occur within 4 weeks after randomization
  Other Names: VT ablation; ischemic VT ablation; catheter ablation; radiofrequency ablation
  Arms: Ablation
Drug: Amiodarone — Amiodarone titrated to therapeutic levels as per standard of care and maintained on a dose of at least 200 mg (300 mg recommended) once a day for the duration of the study
  Other Names: Cordarone
  Arms: Amiodarone

SUMMARY:
Implantable Cardioverter Defibrillators (ICDs) provide a shock or pacing therapy to bring back a normal heart beat when a patient experiences a dangerous abnormal heart rhythm such as ventricular tachycardia (VT). ICDs are very successful in bringing back a normal heart beat when VT occurs, but they do not prevent further dangerous heart rhythms from occurring. This study is designed to determine the best way to manage patients who have an ICD and who continue to have episodes of VT. There are two methods for treatment the VT: 1) Ablation, and 2) Medication.

An ablation procedure involves placing a flexible catheter (insulated wire) in the groin area and threading it into the heart. After the doctor has located the affected area responsible for the VT, radiofrequency energy is delivered by the power generator through the catheter to the inside of the heart. The radiofrequency energy ablates (burns) a small area of the heart tissue thought to cause the VT.

A medication called Amiodarone is an "anti-arrhythmic" prescribed to prevent abnormal heart rhythms from recurring.

The purpose of this study is to compare these two different methods for treating VT. Treatment with ablation and amiodarone are both considered the standard of care for patients with VT but they have not been compared directly in a study like this before.

ELIGIBILITY:
Inclusion Criteria - Patients must meet all of the following criteria:

* > 18 and < 85 years of age
* ICD implanted for primary prophylaxis against sudden cardiac death or ICD implanted for secondary prophylaxis against spontaneous or inducible sustained VT without any reversible causes
* Coronary artery disease (CAD) with prior myocardial infarction (MI)
* ICD or electrocardiogram (ECG) documentation of ventricular arrhythmia responsible for appropriate ICD therapy [antitachycardia pacing (ATP) & shocks].

Exclusion Criteria - Patients should not have any of the following criteria:

* Contraindication or allergy to contrast media, routine procedural medications or catheter materials
* Contraindication to an interventional procedure
* Current or previous (within 3 months) amiodarone therapy
* Atrial Fibrillation requiring antiarrhythmic drug therapy
* Contraindication to amiodarone therapy
* New York Heart Association (NYHA) functional class IV
* Myocardial infarction within the past 60 days
* Stroke within the past 90 days
* Unstable angina
* Hypertrophic cardiomyopathy, Non-ischemic dilated cardiomyopathy, Arrhythmogenic Right Ventricular Dysplasia, Brugada Syndrome, Catecholamine sensitive polymorphic VT or long QT syndrome
* Patients with active ischemia that are eligible for revascularization
* Life expectancy less than 6 months
* Incessant or multiple episodes of VT requiring immediate therapy with medications or ablation
* Untreated hypothyroidism or hyperthyroidism. Patients who are euthyroid on thyroid hormone replacement therapy are acceptable.
* Current enrollment in another investigational drug or device study.
* Presence of any other condition that the investigator feels would be problematic or would restrict or limit the participation of the patient for the entire study period.
* Absolute contra-indication to the use of heparin and or warfarin.
* Documented intra-atrial thrombus, ventricular thrombus (< 6 months after detection of thrombus), tumor, or another abnormality which precludes catheter introduction.
* Females of childbearing potential who are not practicing protocol acceptable method of birth control.

Ages: 19 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, M.D., Principal Investigator — Texas Cardiac Arrhythmia Research Foundation; David J Callans, M.D., Principal Investigator — University of Pennsylvania; Carlos A. Morillo, M.D., Principal Investigator — Population Health Research Institute, McMaster University; Girish M. Nair, M.D., Principal Investigator — Population Health Research Institute, McMaster University
Locations (11):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - University of Virginia Health System, Charlottesville, Virginia
- Canada (5):
  - Hamilton Health Sciences, Hamilton, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - McGill University Health Center, Montreal, Quebec
  - Institut Universitaire de Cardiologie et Pneumologie de Québec, Québec
- Beijng Fuwai Heart Hospital, Beijing, China

REFERENCES:
- See also: Population Health Research Institute — http://www.phri.ca/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ablation | Amiodarone
Started | 7 | 5
Completed | 0 | 0
Not Completed | 7 | 5
Not completed — Study terminated early | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ablation | Amiodarone | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9.7) | 57 (13.4) | 61 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  Canada | 5 | 3 | 8
  United States | 1 | 0 | 1
  China | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Appropriate ICD Therapy, Slow VT or Sudden Cardiac Death
Description: Number of participants with a composite outcome of any of:
  1. Appropriate Implantable Cardioverter Defibrillator (ICD) therapy [Including antitachycardia pacing (ATP) and shocks]
  2. Slow ventricular tachycardia (VT) below ICD detection threshold leading to hospitalization or necessitates antiarrhythmic medications and/or catheter ablation
  3. Sudden Cardiac Death
Time Frame: From 30 days following randomization until final follow-up visit
Measure: Number; unit: participants
Arm/Group | Ablation | Amiodarone
Number analyzed (Participants) | 7 | 5
participants | 1 | 2

2. Secondary Outcome: Number of Participants With (a) Ablation or Amiodarone Complications, (b) Inappropriate Shocks From ICD, or (c) Need for Concomitant Use of Sotalol, Dofetilide, Azimilide or Class 1 Antiarrhythmic Agents in Either Arm of the Trial.
Description: Number of Participants with (a) Ablation or Amiodarone Complications, (b) Inappropriate Shocks from ICD, or (c) Need for Concomitant use of Sotalol, Dofetilide, Azimilide or Class 1 Antiarrhythmic agents in either arm of the trial.
Time Frame: from randomization until final follow-up
Measure: Number; unit: participants
Arm/Group | Ablation | Amiodarone
Number analyzed (Participants) | 7 | 5
participants | 2 | 0

3. Secondary Outcome: Quality of Life Score
Description: Quality of life score in each treatment arm using the EQ-5D Visual Analogue Scale (VAS) (euroqol.org). The EQ-5D VAS is a patient reported scale from 0 to 100 on which the patient rates how good or bad their health is today with 100 being the best health they can imagine and 0 being the worst health they can imagine.
Time Frame: At 6 months follow-up
Population: Participants with data collected at 6 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Ablation | Amiodarone
Number analyzed (Participants) | 3 | 3
score on a scale | 59 [52 to 65] | 83 [70 to 95]

ADVERSE EVENTS:
Time Frame: Follow-up period from date of randomization until final follow-up visit. Events were assessed at 1 month, 6 months and 12 months after randomization.
Description: Note that the study was terminated early for non-feasibility. 12 participants were enrolled, 9 completed 1 month of follow-up, 6 completed 6 months of follow-up and 1 completed 12 months of follow-up.
Arm/Group | Ablation | Amiodarone
Serious Adverse Events (participants affected / at risk) | 2/7 | 1/5
Other Adverse Events (participants affected / at risk) | 0/7 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ablation (N=7) | Amiodarone (N=5)
pneumonia (Infections and infestations) | 0 (0) | 1 (1)
acute renal failure (Renal and urinary disorders) | 0 | 1
pseudo aneurysm (Vascular disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No